CLINICAL TRIAL: NCT04295369
Title: Effect of a Culturally Adapted Self-help Smartphone-based Lifestyle Intervention in Improving Psychological Well-being: A Pilot Randomized Controlled Trial
Brief Title: Lifestyle Hub Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY010
Record Dates: First submitted 2020-02-28; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Psychological Distress
Keywords: Psychological Well-being; Lifestyle Medicine; Self-help; Depression; Anxiety
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Medicine Group (Experimental)
  Interventions: Behavioral: Lifestyle Medicine
- Waitlist Control Group (No Intervention): Participants in the waitlist control group will receive the intervention after the immediate post-treatment assessment.

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Lifestyle intervention with components including physical activity, diet, relaxation/mindfulness, sleep, stress management, and Chinese dietary recommendations.
  Arms: Lifestyle Medicine Group

SUMMARY:
This study will examine the effects of a smartphone-based lifestyle medicine (LM) for improving psychological well-being in Chinese population. Since a range of lifestyle factors are involved in the pathogenesis and progression of common mental disorders (e.g., depression and anxiety), modifying different lifestyle factors simultaneously may be effective to improve our psychological well-being. Chinese dietary recommendations will be integrated into the app to increase the acceptability towards mental health intervention. Through this study, we aim to promote evidence-based patient care and to improve help-seeking and access to evidence-based interventions for improving psychological well-being.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial on the effects of a culturally adapted self-help smartphone-based lifestyle medicine for improving psychological well-being in Chinese population. Prior to all study procedures, eligible participants will be required to complete an online informed consent (with telephone support). Around 30 eligible participants will be randomly assigned to either smartphone-based lifestyle medicine (LM group) or the waitlist control group (WL group) in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged ≥ 18 years
* Able to read Chinese and type in Chinese or English
* Have an Internet-enabled mobile device (iOS or Android operating system)
* Are willing to provide informed consent and comply with the trial protocol

Exclusion Criteria:

* Have a Patient Health Questionnaire (PHQ-9) score ≥ 10
* Have a Generalized Anxiety Disorder 7-Item Scale (GAD-7) ≥ 8
* Current involvement in psychotherapy or unstable medication for depression and/or anxiety
* Beck Depression Inventory (BDI-II) Item 9 score of at least 2 indicating a current moderate suicidal risk that requires active crisis management (referral information to professional services will be provided to those with serious suicidal risk)
* Are having unsafe conditions and are not recommended for physical activity or a change in diet by physicians
* Having major psychiatric, medical or neurocognitive disorders that make participation infeasible or interfere with the adherence to the lifestyle modification

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Depression Anxiety Stress Scales-21 | Immediately post-treatment and 1-month post treatment
  DASS-21 is a 21-items scale, comprises of three sub-scales which measures the negative emotional states of depression, anxiety, and stress, over the past week. The DASS is based on a dimensional rather than a categorical conception of psychological disorder, thus it has no direct implications for the allocation of patients to discrete diagnostic categories. However, recommended cutoff scores for conventional severity labels (normal, moderate, severe) are given in the DASS Manual.

SECONDARY OUTCOMES:
Change in The Insomnia Severity Index (ISI) | Baseline, immediately post-treatment and 1-month post treatment
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5 point Likert scale are obtained on the perceived severity of sleep-onset, sleep maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediately post-treatment and 1-month post treatment
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the Health-Promoting Lifestyle Profile (HPLP II) | Baseline, immediately post-treatment and 1-month post treatment
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
Change in the Sheehan Disability Scale (SDS) | Baseline, immediately post-treatment and 1-month post treatment
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. The participant rates the extent to which work/school, social life and home life or family responsibilities are impaired by his or her symptoms on a 10 point visual analog scale. The numerical ratings of 0-10 can be translated into a percentage, if desired. The 3 items can also be summed into a single dimensional measure of global functional impairment that rages from 0 (unimpaired) to 30 (highly impaired).
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline, immediately post-treatment and 1-month post treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.
Change in the Food Frequency Questionnaires (FFQs) | Baseline, immediately post-treatment and 1-month post treatment
  FFQs is a 18-item scale, including drinks, plant, animal products and cigarette intake, which measures the frequency of food intake over the past three months on a 7-point scale.
Change in the International Physical Activities Questionnaire - Chinese version (IPAQ-C) | Baseline, immediately post-treatment and 1-month post treatment
  Participants' sitting time, walking time and moderate and vigorous physical activity are assessed by 5 questions from a short form of the International Physical Activity Questionnaire - Chinese version.
Self-developed survey | Baseline
  The self-developed survey will collect information including demographic information (e.g., age, gender, level of education, working industry, relationship status, and location of residence), substance use, body mass index (BMI), rest-activity pattern, and social rhythms, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Derived] Wong VW, Tong JT, Shi NK, Ng CH, Sarris J, Ho FY. Smartphone-delivered multicomponent lifestyle medicine intervention for improving mental health in a nonclinical population: a randomized controlled trial. Front Public Health. 2024 Jan 16;11:1231981. doi: 10.3389/fpubh.2023.1231981. eCollection 2023. PMID 38292386